CLINICAL TRIAL: NCT02025283
Title: The Comparison of the Efficacy of Radiofrequency Nucleoplasty and Targeted Disc Decompression in Lumbar Radiculopathy: A Retrospective Review
Brief Title: Efficacy of Radiofrequency Nucleoplasty and Targeted Disc Decompression in Lumbar Radiculopathy
Acronym: RFNaTDD
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Barıs Adaklı, Specialist, Ankara University
Other Study IDs: 10-402-13
Record Dates: First submitted 2013-12-24; First posted 2014-01-01 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Visual Analogue Pain Scale; Pain Measurement
Keywords: Intervertebral disc disease; Radiculopathy; Chronic pain; Thermocoagulation
MeSH Terms: conditions — Intervertebral disc disease; Radiculopathy; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group Decompression: Group Decompression: Patients assigned to Group Decompression. After determination of the appropriate space for the approach under fluoroscopy guidance, a 17 gauge trochar needle was advanced posterolaterally up to the center of the disc. Then site verification was done again with water soluble contrast material under floroscopy guidance. Then flexible intradiscal decompression catheter (SpineCATH®, Smith & Nephew, Memphis, TN) were advanced inside the trochar needle towards the disc and decompression was performed. After being sure of achieving sufficient decompression inside the disc, the decompression device were removed under fluoroscopy guidance and the incision site was closed and the patients were recommended to have bedrest for 2 hours.
  Interventions: Procedure: Group Decompression or Group Nucleoplasty
- Group Nucleoplasty: Group Nucleoplasty : Patients assigned to Group Nucleoplasty. After determination of the appropriate space for the approach under fluoroscopy guidance, a 17 gauge trochar needle was advanced posterolaterally up to the center of the disc. Then site verification was done again with water soluble contrast material under floroscopy guidance. Then radiofrequency-compatible needle (Coblation: Perc DLE SpineWandTM [ArthroCare Spine, Sunnyvale, CA] were advanced inside the trochar needle towards the disc and nucleoplasty was performed. After being sure of achieving sufficient decompression inside the disc, the nucleoplasty probe was removed under fluoroscopy guidance and the incision site was closed and the patients were recommended to have bedrest for 2 hours.
  Interventions: Procedure: Group Decompression or Group Nucleoplasty

INTERVENTIONS:
Procedure: Group Decompression or Group Nucleoplasty — Group Decompression: Decompression with flexible intradiscal decompression catheter (SpineCATH®, Smith & Nephew, Memphis, TN) Group Nucleoplasty: Nucleoplasty with radiofrequency-compatible needle (Coblation: Perc DLE SpineWandTM [ArthroCare Spine, Sunnyvale, CA]
  Other Names: ArthroCare Spine; SpineCATH®

SUMMARY:
The aim of this study is to compare early and long term efficacy of lumbar radiofrequency nucleoplasty and targeted disc decompression in patients with lumbar radiculopathy who failed previous conventional therapy. Medical records of 37 patients undergoing targeted disc decompression, 36 patients undergoing lumbar radiofrequency nucleoplasty were retrospectively examined.Visual Analogue Scale (VAS), Numerical Rating Scale (NRS), Functional Rating Index, Backache index, Oswestry Lumbar Back Pain Disability Index, Rolland-Morris Lumbar Back Pain Questionnaire scales were used before treatment and 1,6,12 months after the procedure. North American Spine Society Satisfaction Scale was used at 12th month after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* patients having radicular pain with or without low back pain for at least 6 weeks inspite of conservative treatment who have unsequestrated, bulging, protruded or extruded hernia confirmed with MRI.

Exclusion Criteria:

* patients having a more than 50% loss in disc area, sequestrated disc, the presence of vertebra fracture or tumor, the patients having spinal stenosis or spondylolisthesis

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 120 patients with lumbar radiculopathy undergoing nucleoplasty and targetted disc decompression in Algology Department of a University Hospital between 2010 and 2012 were retrospectively evaluated and complete data of only 73 patients were reached and they were included to the study
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Decrease in Visual Analogue Scale (VAS) | 12 months

SECONDARY OUTCOMES:
More than 50% procedure-related patient satisfaction ratio in North American Spine Society Satisfaction Scale | 12 months

OTHER OUTCOMES:
Decrease in Numerical Rating Scale | 12 months
Decrease in Functional Rating Index | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Barış Adaklı, Specialist, Principal Investigator — Ankara University
Locations (1):
- Ankara University Medical School Algology Department, Ankara, Turkey (Türkiye)